CLINICAL TRIAL: NCT00625573
Title: Phase II Trial of Abraxane and Capecitabine in Metastatic Colon Cancer (COL 01)
Acronym: ABX067
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mt. Sinai Medical Center, Miami (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Joseph Pizzolato, M.D., Mt. Sinai Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: COL-01
Record Dates: First submitted 2008-02-19; First posted 2008-02-28 (Estimated); Last update posted 2009-09-18 (Estimated); Status verified 2009-09

CONDITIONS: Colorectal Cancer
Keywords: Colon Cancer; Abraxis Oncology; Abraxane; Phase II; Colorectal; Mt. Sinai Medical Center; CCOP
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms | interventions — Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Abraxane — 100mg/m2 every week X's 3

SUMMARY:
This is an open-label, phase II study to evaluate the efficacy and safety of Abraxane in combination with Capecitabine in patients with metastatic colorectal cancer in the second or third line

DETAILED DESCRIPTION:
Inclusion Criteria

* Signed written informed consent
* Patients with histologically or cytologically confirmed stage IV colorectal cancer who have failed either irinotecan-based, oxaliplatin-based or both. ECOG performance status of 0-2
* Presence of measurable disease by radiographic study (including CT or MRI scan, or chest x-ray) or physical examination
* At least 3 weeks since last major surgery.
* At least 6 weeks since prior radiotherapy providing that the extent and site of radiotherapy fields are such that marked bone marrow suppression is NOT expected. Patients who have received palliative radiotherapy must have recovered from any reversible toxic effects e.g. nausea and vomiting caused by radiation of fields.
* At least 4 weeks since prior chemotherapy.
* Pt with reproductive potential must use effective BC

Required Screening Laboratory Criteria:

* Hemoglobin 9.0g/dL
* WBC 3,500/mm3 [ 3.5 x 109/L]
* Neutrophils 1,500/mm3 [1.5 x 109/L]
* Platelets 100,000/mm3 [ 100.0 x 109/L]
* Creatinine 1.5 mg/dL (133 micromol/L) AND creatinine clearance 60 mL/min • A probable life expectancy of at least 6 months.

Exclusion Criteria

* No brain metastases.
* If female of childbearing potential, pregnancy test is negative.
* Concomitant malignancies or previous malignancies other than colorectal cancer within the last five years, with the exception of adequately treated basal or squamous cell carcinoma of the skin, carcinoma in situ of the cervix, or low grade prostate cancer.
* Active infection.
* Concurrent severe medical problems unrelated to the malignancy, which would significantly limit full compliance with the study or expose the patient to extreme risk.
* Sexually active patients refusing to practice adequate contraception. (condom plus spermicide, or other form of birth control)
* Patients with conditions which might affect absorption of an oral drug (for example intermittent obstruction) should be excluded unless discussed and agreed with the principal investigator
* History of grade 3 or 4 toxicity to fluoropyrimidines.
* Pre-existing neuropathy ≥ NCI CTC grade 2

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* Patients with histologically or cytologically confirmed stage IV colorectal cancer who have failed either irinotecan-based, oxaliplatin-based or both. ECOG performance status of 0-2
* Presence of measurable disease by radiographic study (including CT or MRI scan, or chest x-ray) or physical examination
* At least 3 weeks since last major surgery.
* At least 6 weeks since prior radiotherapy providing that the extent and site of radiotherapy fields are such that marked bone marrow suppression is NOT expected. Patients who have received palliative radiotherapy must have recovered from any reversible toxic effects e.g. nausea and vomiting caused by radiation of fields.
* At least 4 weeks since prior chemotherapy.
* Pt with reproductive potential must use effective BC
* Required Screening Laboratory Criteria:

  * Hemoglobin 9.0g/dL
  * WBC 3,500/mm3 [ 3.5 x 109/L]
  * Neutrophils 1,500/mm3 [1.5 x 109/L]
  * Platelets 100,000/mm3 [ 100.0 x 109/L]
  * Creatinine 1.5 mg/dL (133 micromol/L) AND creatinine clearance 60 mL/min
* A probable life expectancy of at least 6 months

Exclusion Criteria:

* No brain metastases.
* If female of childbearing potential, pregnancy test is negative.
* Concomitant malignancies or previous malignancies other than colorectal cancer within the last five years, with the exception of adequately treated basal or squamous cell carcinoma of the skin, carcinoma in situ of the cervix, or low grade prostate cancer.
* Active infection.
* Concurrent severe medical problems unrelated to the malignancy, which would significantly limit full compliance with the study or expose the patient to extreme risk.
* Sexually active patients refusing to practice adequate contraception. (condom plus spermicide, or other form of birth control)
* Patients with conditions which might affect absorption of an oral drug (for example intermittent obstruction) should be excluded unless discussed and agreed with the principal investigator
* History of grade 3 or 4 toxicity to fluoropyrimidines.
* Pre-existing neuropathy ≥ NCI CTC grade 2.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2007-09; Primary Completion 2009-02 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
To evaluate the efficacy by means of response rate of Abraxane and capecitabine in combination, in the treatment of patients with colorectal cancer in the 2nd or 3rd line metastatic setting following failure of irinotecan or oxaliplatin based therapy | One year

SECONDARY OUTCOMES:
To evaluate overall survival, time to progression, response duration, time to response and safety of this combination | One Year

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Pizzolato, MD, Principal Investigator — Mt. Sinai Medical Center Miami Beach Florida
Locations (1):
- Mount Sinai Medical Center, Miami Beach, Florida, United States